CLINICAL TRIAL: NCT03581474
Title: Evaluation of a Bronchoalveolar Lavage Procedure With a Flexible Disposable Bronchoscope, Ambu aScope 3 Large in Patients in an Intensive Care Unit Setting
Brief Title: Evaluation of BAL Procedure With Ambu aScope 3 Large in Patients in an ICU Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Ambu A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIS-001
Record Dates: First submitted 2017-09-22; First posted 2018-07-10 (Actual); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2018-06

CONDITIONS: Atelectasis; Bronchoscopy
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- aScope 3 Large (Other): Bronchoscopic procedure
  Interventions: Device: Bronchoscopic procedure

INTERVENTIONS:
Device: Bronchoscopic procedure — Single-use flexible bronchoscope aScope 3 Large

SUMMARY:
An Investigation to determine the single-use scope's ability to suction secretion from the lungs to resolve the collapse of the lung.

DETAILED DESCRIPTION:
The purpose of this investigation it to determine the single-use scope's ability to suction secretion from the lungs to resolve the collapse of the lung. The hypothesis is that aScope 3 Large is able to manage the secretion and thereby facilitating the resolution of secretion in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Clinical indication and eligible for a BAL procedure, as judged by the investigator
* Patients being admitted in the ICU at the investigational centre
* Provision of signed IC by subject, or subject's legal representative e.g. next of kin

Exclusion Criteria:

* Patients where BAL treatment cannot be clinically justified, judged by the investigator
* ETT >7 mm and ≤8.5 mm in diameter
* Participating in other interventional clinical investigations or have previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Charlotte Lundgaard, Study Chair — Ambu A/S
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | aScope 3 Large
Started | 12
Completed (Early completion due to recruitment issues. Originally the study aimed to include 90 subjects.) | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | aScope 3 Large
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 173.9 (10.2)
Weight [Mean (Standard Deviation); unit: kg] | 113.3 (39.3)
ASA-score [Count of Participants; unit: Participants] — I. Patient is a completely healthy fit patient. II. Patient has mild systemic disease. III. Patient has severe systemic disease that is not incapacitating. IV. Patient has incapacitating disease that is a constant threat to life. V. A moribund patient who is not expected to live 24 hour with or without surgery.
  Participants
    I. | 0
    II. | 5
    III. | 6
    IV. | 1
    V. | 0
Indication for invasive mechanical ventilation [Count of Participants; unit: Participants]
  Cardiogenic shock | 4
  Lung transplant | 1
  Respiratory failure | 4
  Cardiac arrest | 1
  Severe aortic stenosis | 1
  aortic regurgitation | 1
Endotracheal tube size [Count of Participants; unit: Participants]
  Size 7 | 1
  Size 7.5 | 4
  Size 8 | 6
  Size 8.5 | 1

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Oxygenation (PaO2/FiO2 Ratio) After a BAL Treatment
Description: Resolution of atelectasis measured by improvement in oxygenation after a bronchoscopic procedure (bronchoalveolar lavage treatment). PaO2/FiO2 ratio will be compared between baseline and 4 hourst post the BAL procedure.
Time Frame: 4 hours after procedure
Population: Missing data at 4h post measures for one subject
Measure: Mean (Standard Deviation); unit: PaO2/FiO2
Arm/Group | aScope 3 Large
Number analyzed (Participants) | 12
PaO2/FiO2
  PaO2/FiO2 Baseline: number analyzed (Participants) | 11
  PaO2/FiO2 Baseline | 194.69 (111.27)
  PaO2/FiO2 4h post | 211.54 (94.92)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 4 hours post procedure
Arm/Group | aScope 3 Large
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03581474/Prot_SAP_000.pdf